CLINICAL TRIAL: NCT02032017
Title: Percutaneous Assisted Approach for Total Hip Replacement and it's Effect on Functional Rehabilitation Compared to the Anterolateral Approach.
Brief Title: Percutaneous Assisted Approach for Total Hip Replacement and it's Effect on Functional Rehabilitation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Stöpler Belgium nv (Unknown)
Responsible Party: Principal Investigator, Claudia Hendrickx, PhD student, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B300201318915
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Total Hip Arthroplasty
Keywords: Total Hip Arthroplasty; Gluteus medius; Approach; Rehabilitation; Functional outcome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous assisted approach (Experimental): In this technique, a second small incision (1 cm) at the anterior border of the femur is made. A canulla is placed underneath the muscle and used to pass the reamers in the direction of the acetabulum. There's no need to enlarge the skin incision or to release more muscle insertion to achieve good working access to the acetabulum. Two advantages can be defined: sparing of the gluteus medius muscle and safe access to the acetabulum to obtain perfect positioning of the implants.
  Interventions: Procedure: Ceramic on ceramic couple; Procedure: Percutaneous assisted approach; Other: Usual care
- Anterolateral approach (Active Comparator): A standard transgluteal approach is used. This means a large part of the gluteus medius muscle is released to obtain good access to the acetabulum.
  Interventions: Procedure: Ceramic on ceramic couple; Procedure: Anterolateral approach; Other: Usual care

INTERVENTIONS:
Procedure: Ceramic on ceramic couple — All patients will get a standard total hip replacement (cementless hydroxyapatite coated cup and a titanium plasmasprayed stem) with a ceramic on ceramic (third generation biolox delta) couple. Preoperative leg length and offset are marked to reconstruct the preoperative leg length and to obtain the optimal offset.
Procedure: Percutaneous assisted approach
  Arms: Percutaneous assisted approach
Procedure: Anterolateral approach
  Arms: Anterolateral approach
Other: Usual care — Both groups will receive usual care (UC) after surgery. This includes standard physiotherapy care consisting of mobilizing and strengthening techniques. All patients will receive a booklet containing information about the surgery, weight bearing after the surgery, and rehabilitation in general.

SUMMARY:
The purpose of this study is to investigate whether revalidation following total hip replacement through the percutaneous approach is faster or better than following the anterolateral approach. We assume this would be the case since it is possible to spare a large part of the gluteus medius muscle with the percutaneous approach.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hip arthritis or avascular necrosis (AVN) in need for total hip replacement

Exclusion Criteria:

* Comorbidities affecting functional outcome
* Symptomatic lumbar pathology
* Need of surgery or intervention on the ipsilateral knee and/or ankle/foot
* Neurological disorders such as Parkinsonism and previous cardiovascular accidents (CVA)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
change in time needed for the timed get up and go test | baseline, 4 weeks, 12 weeks
  The subject is asked to stand up from a chair, walk 3m to a cone, return to the chair and sit down again. The time needed to perform this test is recorded in seconds.

SECONDARY OUTCOMES:
surface electromyography (sEMG) of gluteus medius | baseline
  sEMG of the gluteus medius is recorded during maximally voluntary isometric contraction and during single leg stance.
Change in hip abductor muscle strength measured by MicroFET 2 | baseline, 4 weeks, 12 weeks
  The patient lies supine. Resistance is administered on the lateral side of the leg, just proximal of the knee joint. Patients will be asked for a maximally voluntary isometric contraction. The test will be repeated 3 times. The mean value will be recorded.
Change in knee extensor muscle strength measured by MicroFET 2 | baseline, 4 weeks, 12 weeks
  The patient is seated with the hips and knees bent 90°. Resistance is administered on the ventral side of the leg, just proximal of the ankle joint. Patients will be asked for a maximally voluntary isometric contraction. The test will be repeated 3 times. The mean value will be recorded.
Score on the Trendelenburg test | baseline
  The patient is asked to raise one leg (sound side) and lift the non-stance side of the pelvis as high as possible for 30 seconds. The response is classified as followed:
  1. Normal: the pelvis on the non-stance side can be lifted maximally during 30 seconds
  2. The pelvis on the non-stance side can be lifted, but not maximally
  3. The pelvis on the non-stance side is elevated, but not maintained for 30 seconds.
  4. No elevating of the pelvis on the non-stance side
  5. Drooping of the pelvis
  6. Non-valid response: due to hip pain or uncooperative patient
Change in score on the Oxford Hip Score | baseline, 4 weeks, 12 weeks
  The Oxford Hip Score (OHS) is a disease-specific questionnaire that consists of 12 questions for the evaluation of pain and hip function in relation to various activities. Each question contains 5 quantifiable answers, leading to a total score that can range from 12 (least problems) to 60 (most problems).
Change in score on the SF-36 and it's subscales | baseline, 4 weeks, 6 weeks
  The SF-36 is a generic questionnaire that contains 36 items measuring health on 8 different dimensions. These dimensions cover functional status, wellbeing and overall evaluation of health.
Change in time needed to complete the 5 times sit-to-stand test | baseline, 4 weeks, 12 weeks
  This easily feasible test where the patient has to stand up and sit back down 5 times as fast as possible is a good predictor of falling. A worse score (i.e. a longer time needed to complete the test) on the 5 times sit to stand (5tSTS) implies a greater chance of falling.
Change in distance walked during the 6 minute walking test | baseline, 4 weeks, 12 weeks
  The test measures the distance a patient can quickly walk on a flat, hard surface in a time-period of 6 minutes.
surface electromyography (sEMG) of gluteus medius | 4 weeks
  sEMG of the gluteus medius is recorded during maximally voluntary isometric contraction and during single leg stance.
surface electromyography (sEMG) of gluteus medius | 12 weeks
  sEMG of the gluteus medius is recorded during maximally voluntary isometric contraction and during single leg stance.
Score on the trendelenburg test | 4 weeks
  The patient is asked to raise one leg (sound side) and lift the non-stance side of the pelvis as high as possible for 30 seconds. The response is classified as followed:
  1. Normal: the pelvis on the non-stance side can be lifted maximally during 30 seconds
  2. The pelvis on the non-stance side can be lifted, but not maximally
  3. The pelvis on the non-stance side is elevated, but not maintained for 30 seconds.
  4. No elevating of the pelvis on the non-stance side
  5. Drooping of the pelvis
  6. Non-valid response: due to hip pain or uncooperative patient
Score on the Trendelenburg test | 12 weeks
  The patient is asked to raise one leg (sound side) and lift the non-stance side of the pelvis as high as possible for 30 seconds. The response is classified as followed:
  1. Normal: the pelvis on the non-stance side can be lifted maximally during 30 seconds
  2. The pelvis on the non-stance side can be lifted, but not maximally
  3. The pelvis on the non-stance side is elevated, but not maintained for 30 seconds.
  4. No elevating of the pelvis on the non-stance side
  5. Drooping of the pelvis
  6. Non-valid response: due to hip pain or uncooperative patient

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Hendrickx, PhD student, Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - UZA, Antwerp, Antwerp
  - ZNA Middelheim, Wilrijk, Antwerp

REFERENCES:
- [Derived] Hendrickx C, De Hertogh W, Van Daele U, Mertens P, Stassijns G. Effect of percutaneous assisted approach on functional rehabilitation for total hip replacement compared to anterolateral approach: study protocol for a randomized controlled trial. Trials. 2014 Oct 8;15:392. doi: 10.1186/1745-6215-15-392. PMID 25298243